CLINICAL TRIAL: NCT04707313
Title: A PHASE 2B, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL GROUP, DOSE-RANGING STUDY TO EVALUATE THE EFFICACY AND SAFETY OF PF-06882961 ADMINISTRATION IN ADULTS WITH OBESITY
Brief Title: A Study to Evaluate the Efficacy and Safety of PF-06882961 in Adults With Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3421019; 2020-001312-19 (EudraCT Number)
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: Weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — danuglipron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Placebo (Cohorts 1 and 2) (Placebo Comparator)
  Interventions: Drug: Placebo (Cohorts 1 and 2)
- PF-06882961 40 milligrams (mg) twice daily (BID), 1-week titration (Cohort 1) (Experimental): The dose will be titrated with 1 week of dosing at each step to reach the target dose of 40 mg BID.
  Interventions: Drug: PF-06882961 (Cohorts 1 and 2)
- PF-06882961 80 mg BID, 1-week titration (Cohort 1) (Experimental): The dose will be titrated with 1 week of dosing at each step to reach the target dose of 80 mg BID.
  Interventions: Drug: PF-06882961 (Cohorts 1 and 2)
- PF-06882961 120 mg BID, 1-week titration (Cohort 1) (Experimental): The dose will be titrated with 1 week of dosing at each step to reach the target dose of 120 mg BID.
  Interventions: Drug: PF-06882961 (Cohorts 1 and 2)
- PF-06882961 160 mg BID, 1-week titration (Cohort 1) (Experimental): The dose will be titrated with 1 week of dosing at each step to reach the target dose of 160 mg BID.
  Interventions: Drug: PF-06882961 (Cohorts 1 and 2)
- PF-06882961 200 mg BID, 1-week titration (Cohort 1) (Experimental): The dose will be titrated with 1 week of dosing at each step to reach the target dose of 200 mg BID.
  Interventions: Drug: PF-06882961 (Cohorts 1 and 2)
- PF-06882961 120 mg BID, 2-week titration (Cohorts 1 and 2) (Experimental): The dose will be titrated with 2 weeks of dosing at each step to reach the target dose of 120 mg BID.
  Interventions: Drug: PF-06882961 (Cohorts 1 and 2)
- PF-06882961 160 mg BID, 2-week titration (Cohorts 1 and 2) (Experimental): The dose will be titrated with 2 weeks of dosing at each step to reach the target dose of 160 mg BID.
  Interventions: Drug: PF-06882961 (Cohorts 1 and 2)
- PF-06882961 200 mg BID, 2-week titration (Cohorts 1 and 2) (Experimental): The dose will be titrated with 2 weeks of dosing at each step to reach the target dose of 200 mg BID.
  Interventions: Drug: PF-06882961 (Cohorts 1 and 2)
- Placebo (Cohort 3) (Placebo Comparator)
  Interventions: Drug: Placebo (Cohort 3)
- PF-06882961 80 mg BID, 4-week titration (Cohort 3) (Experimental): The dose will be titrated with 4 weeks of dosing at each step to reach the target dose of 80 mg BID.
  Interventions: Drug: PF-06882961 (Cohort 3)
- PF-06882961 140 mg BID, 4-week titration (Cohort 3) (Experimental): The dose will be titrated with 4 weeks of dosing at each step to reach the target dose of 140 mg BID.
  Interventions: Drug: PF-06882961 (Cohort 3)
- PF-06882961 200 mg BID, 4-week titration (Cohort 3) (Experimental): The dose will be titrated with 4 weeks of dosing at each step to reach the target dose of 200 mg BID.
  Interventions: Drug: PF-06882961 (Cohort 3)

INTERVENTIONS:
Drug: Placebo (Cohorts 1 and 2) — 4 matching placebo tablets taken twice daily
  Arms: Placebo (Cohorts 1 and 2)
Drug: PF-06882961 (Cohorts 1 and 2) — Participants will be randomized to one of 5 active target dose levels (40, 80, 120, 160 or 200 mg BID) achieved through 1-week titration steps, or 3 active target dose levels (120, 160 or 200 mg BID) achieved through 2-week titration steps, taking 4 tablets twice daily
  Arms: PF-06882961 120 mg BID, 1-week titration (Cohort 1); PF-06882961 120 mg BID, 2-week titration (Cohorts 1 and 2); PF-06882961 160 mg BID, 1-week titration (Cohort 1); PF-06882961 160 mg BID, 2-week titration (Cohorts 1 and 2); PF-06882961 200 mg BID, 1-week titration (Cohort 1); PF-06882961 200 mg BID, 2-week titration (Cohorts 1 and 2); PF-06882961 40 milligrams (mg) twice daily (BID), 1-week titration (Cohort 1); PF-06882961 80 mg BID, 1-week titration (Cohort 1)
Drug: Placebo (Cohort 3) — 2 matching placebo tablets taken twice daily
  Arms: Placebo (Cohort 3)
Drug: PF-06882961 (Cohort 3) — Participants will be randomized to one of 3 active target dose levels (80, 140 or 200 mg BID) achieved through 4-week titration steps, taking 2 tablets twice daily.
  Arms: PF-06882961 140 mg BID, 4-week titration (Cohort 3); PF-06882961 200 mg BID, 4-week titration (Cohort 3); PF-06882961 80 mg BID, 4-week titration (Cohort 3)

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called PF-06882961) for the potential treatment of obesity. The study will compare the experiences of participants taking the study medicine (PF-06882961) to those of participants who take placebo (a look- alike substance that contains no active study medicine). The aim is to measure the body's response to the study medicine, including any changes in participants' body weight, waist and hip measurements, how well they tolerate the study medicine, and to measure levels of the study medicine in participants' blood.

This study is seeking participants who have obesity, who do not have diabetes and who have had a stable body weight and not participated in a formal weight loss program in the 90 days before the study. The study medicine or placebo will be taken as tablets by mouth 2 times a day (1 time in the morning and 1 time in the evening).

There are 3 groups of participants (called cohorts) in this study. For participants in Cohorts 1 and 2, total study participation will be about 9 months, with 15 planned study visits (14 visits to the study clinic and 1 telephone call). For participants in Cohort 3, total study participation will be about 10 months, with 21 planned study visits (12 visits to the study clinic and 9 telephone calls).

ELIGIBILITY:
Inclusion Criteria:

* Participants with obesity, defined as a Body Mass Index greater than or equal to 30.0 kg/m2
* Stable body weight, defined as <5 kg change (per participant report) for 90 days before visit 1

Exclusion Criteria:

* Any condition possibly affecting drug absorption
* Current or prior diagnosis of Type 1 or Type 2 diabetes mellitus or secondary forms of diabetes
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, heart failure, or transient ischemic attack within 6 months prior to visit 1
* Any malignancy not considered cured
* Personal or family history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 or suspected MTC
* History of acute pancreatitis within 180 days (6 months) prior to visit 1 or any history of chronic pancreatitis
* Symptomatic gallbladder disease
* Medical history or characteristics suggestive of genetic or syndromic obesity or obesity induced by other endocrinological disorders
* History of major depressive disorder or other severe psychiatric disorders within the last 2 years
* Any lifetime history of a suicide attempt
* Known medical history of active liver disease, including chronic active hepatitis B or C, or primary biliary cirrhosis
* Known history of HIV
* Supine blood pressure greater than or equal to 160 mmHg (systolic) or greater than or equal to 100 mmHg (diastolic)
* Clinically relevant ECG abnormalities
* Positive urine drug screen
* Participation in a formal weight reduction program within 90 days prior to visit 1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- United States (27):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Velocity Clinical Research - Westlake, Los Angeles, California
  - Alliance for Multispecialty Research, LLC, Coral Gables, Florida
  - Optimus U Corporation, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Clinical Investigation Specialists, Gurnee, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Velocity Clinical Research, Valparaiso, Valparaiso, Indiana
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - ActivMed Practices & Research, LLC, Methuen, Massachusetts
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Velocity Clinical Research, Inc., Cleveland, Ohio
  - Clinical Trials of South Carolina, Moncks Corner, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Palmetto Primary Care Physicians (Sub-I physicals only), Summerville, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - PMG Research, Inc. d/b/a PMG Research of Knoxville, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
- Canada (8):
  - Rivergrove Medical Clinic, Winnipeg, Manitoba
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Milestone Research , Inc, London, Ontario
  - Manna Research Toronto, Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Alpha Recherche Clinique, Québec, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
  - Centre de Recherche Saint-Louis, Québec
- Japan (4):
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Tokyo Center Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Medical Corporation Heishinkai ToCROM Clinic, Shinjuku-ku, Tokyo
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Buckeridge C, Cobain S, Bays HE, Matsuoka O, Fukushima Y, Halstead P, Tsamandouras N, Sherry N, Gorman DN, Saxena AR. Efficacy and safety of danuglipron (PF-06882961) in adults with obesity: A randomized, placebo-controlled, dose-ranging phase 2b study. Diabetes Obes Metab. 2025 Sep;27(9):4915-4926. doi: 10.1111/dom.16534. Epub 2025 Jun 20. PMID 40539310
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421019

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1220 participants were screened (Cohorts 1 and 2: 926 and Cohort 3: 294), of which 592 failed screening and 628 were randomized (Cohorts 1 and 2: 499 and Cohort 3: 129) in the study. Data for participants with the same dose and dosing frequency from Cohorts 1 and 2 were combined as pre-specified in the statistical analysis plan.
Groups:
- Cohorts 1 and 2: Placebo: Participants received placebo matched to PF-06882961 twice daily (BID), orally for a total of 26 weeks.
- Cohort 1: PF-06882961 40 mg BID (1-week Titration): Participants received oral daily doses of PF-06882961, titrated with 1-week at each step to a target dose of 40 mg BID, for a total of 26 weeks.
- Cohort 1: PF-06882961 80mg BID (1-week Titration): Participants received oral daily doses of PF-06882961, titrated with 1-week at each step to a target dose of 80 mg BID, for a total of 26 weeks.
- Cohort 1: PF-06882961 120mg BID (1-week Titration): Participants received oral daily doses of PF-06882961, titrated with 1-week at each step to a target dose of 120 mg BID, for a total of 26 weeks.
- Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration): Participants received oral daily doses of PF-06882961, titrated with 2-week at each step to a target dose of 120 mg BID, for a total of 26 weeks.
- Cohort 1: PF-06882961 160 mg BID (1-week Titration): Participants received oral daily doses of PF-06882961, titrated with 1-week at each step to a target dose of 160 mg BID, for a total of 26 weeks.
- Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration): Participants received oral daily doses of PF-06882961, titrated with 2-week at each step to a target dose of 160 mg BID, for a total of 26 weeks.
- Cohort 1: PF-06882961 200 mg BID (1-week Titration): Participants received oral daily doses of PF-06882961, titrated with 1-week at each step to a target dose of 200 mg BID, for a total of 26 weeks.
- Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration): Participants received oral daily doses of PF-06882961, titrated with 2-week at each step to a target dose of 200 mg BID, for a total of 26 weeks.
- Cohort 3: Placebo: Participants received placebo matched to PF-06882961 BID, orally for 32 weeks.
- Cohort 3: PF-06882961 80mg BID (4-week Titration): Participants received oral daily doses of PF-06882961, titrated with 4-week at each step to a target dose of 80 mg BID, for 32 weeks.
- Cohort 3: PF-06882961 140mg BID (4-week Titration): Participants received oral daily doses of PF-06882961, titrated with 4-week at each step to a target dose of 140 mg BID, for 32 weeks.
- Cohort 3: PF-06882961 200mg BID (4-week Titration): Participants received oral daily doses of PF-06882961, titrated with 4-week at each step to a target dose of 200 mg BID, for 32 weeks.
Period: Cohorts 1 and 2(Week 1 - Week 26)
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40 mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration) | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Started | 71 | 62 | 64 | 64 | 38 | 63 | 37 | 64 | 36 | 0 | 0 | 0 | 0
Received Treatment | 71 | 62 | 63 | 64 | 38 | 63 | 37 | 63 | 36 | 0 | 0 | 0 | 0
Completed | 44 | 27 | 30 | 26 | 13 | 18 | 11 | 14 | 13 | 0 | 0 | 0 | 0
Not Completed | 27 | 35 | 34 | 38 | 25 | 45 | 26 | 50 | 23 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 20 | 23 | 25 | 15 | 38 | 15 | 42 | 16 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 5 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 4 | 4 | 5 | 3 | 2 | 3 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 4 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 5 | 3 | 7 | 3 | 4 | 6 | 4 | 4 | 0 | 0 | 0 | 0
Not completed — Randomized not treated | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Cohort 3 (Week 0 to Week 32)
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40 mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration) | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 (Participants who were randomized to Cohort 3 of the study.) | 37 (Participants who were randomized to Cohort 3 of the study.) | 37 (Participants who were randomized to Cohort 3 of the study.) | 36 (Participants who were randomized to Cohort 3 of the study.)
Received Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 37 | 37 | 36
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 13 | 15 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 24 | 22 | 25
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 16 | 18
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 2 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40 mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration) | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration) | Total
Number analyzed (Participants) | 71 | 62 | 63 | 64 | 38 | 63 | 37 | 63 | 36 | 19 | 37 | 37 | 36 | 626
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 28 | 27 | 26 | 21 | 14 | 22 | 17 | 25 | 11 | 8 | 12 | 13 | 14 | 238
  45-64 years | 34 | 31 | 30 | 36 | 17 | 34 | 20 | 31 | 20 | 9 | 24 | 24 | 19 | 329
  Greater than or equal to (>=)65 years | 9 | 4 | 7 | 7 | 7 | 7 | 0 | 7 | 5 | 2 | 1 | 0 | 3 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 40 | 41 | 42 | 22 | 41 | 22 | 41 | 23 | 12 | 23 | 23 | 22 | 397
  Male | 26 | 22 | 22 | 22 | 16 | 22 | 15 | 22 | 13 | 7 | 14 | 14 | 14 | 229
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 8 | 7 | 3 | 2 | 4 | 2 | 5 | 0 | 2 | 3 | 2 | 51
  Not Hispanic or Latino | 65 | 55 | 54 | 56 | 34 | 61 | 33 | 60 | 30 | 19 | 34 | 34 | 34 | 569
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
  Asian | 11 | 8 | 10 | 8 | 3 | 10 | 2 | 13 | 2 | 0 | 0 | 0 | 0 | 67
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 4 | 4 | 10 | 11 | 4 | 8 | 5 | 5 | 3 | 3 | 8 | 6 | 5 | 76
  White | 55 | 48 | 42 | 45 | 31 | 42 | 30 | 45 | 31 | 16 | 29 | 31 | 28 | 473
  More than one race | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Cohorts 1 and 2: Percent Change From Baseline in Body Weight at End of Treatment at Week 26
Description: Percent change from baseline in body weight at end of treatment was reported in this outcome measure. Analysis was performed using MMRM with treatment, time, strata (females versus males) and treatment-by-time interaction as fixed effects, natural log-transformed baseline as a covariate and the (natural log-transformed baseline)-by-time interaction with time fitted as a repeated effect and participant as a random effect. Values were back-transformed from the log scale. Percent change = 100 multiply by [*](back-transformed LS Mean minus [-] 1). Baseline was defined as the average of the duplicate measurements collected closest prior to dosing at Day 1.
Time Frame: Baseline, Week 26
Population: Estimand Set 1 included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Cohort 1: PF-06882961 40mg BID (1-week Titration): Participants received oral daily doses of PF-06882961, titrated with 1-week at each step to a target dose of 40 mg BID, for a total of 26 weeks.
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 71 | 62 | 63 | 64 | 38 | 63 | 37 | 63 | 36
Percent change | 0.17 (0.008) | -5.43 (0.009) | -4.83 (0.009) | -8.94 (0.009) | -6.43 (0.012) | -9.36 (0.010) | -6.96 (0.013) | -8.96 (0.011) | -7.02 (0.012)
Statistical Analysis 1: Comparison: Cohorts 1 and 2: Placebo vs Cohort 1: PF-06882961 40mg BID (1-week Titration); Test type: Superiority; p < .0001, Mixed Models Analysis; Difference to placebo = -5.60, 90% CI 2-sided [-7.41 to -3.74], Standard Error of Mean 0.012 — MMRM:treatment,time,strata(female vs male),treatment-by-time interaction as fixed effect, natural log-transformed baseline as covariate,natural log-transformed baseline-by-time interaction with time fitted:repeated effect, participant:random effect
Statistical Analysis 2: Comparison: Cohorts 1 and 2: Placebo vs Cohort 1: PF-06882961 80mg BID (1-week Titration); Test type: Superiority; p < .0001, Mixed Models Analysis; Difference to placebo = -5.00, 90% CI 2-sided [-6.80 to -3.16], Standard Error of Mean 0.012 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohorts 1 and 2: Placebo vs Cohort 1: PF-06882961 120mg BID (1-week Titration); Test type: Superiority; p < .0001, Mixed Models Analysis; Difference to Placebo = -9.10, 90% CI 2-sided [-10.89 to -7.28], Standard Error of Mean 0.012 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration); Test type: Superiority; p < .0001, Mixed Models Analysis; Difference to Placebo = -6.60, 90% CI 2-sided [-8.75 to -4.39], Standard Error of Mean 0.014 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Cohort 1: PF-06882961 160 mg BID (1-week Titration); Test type: Superiority; p < .0001, Mixed Models Analysis; Difference to Placebo = -9.52, 90% CI 2-sided [-11.43 to -7.56], Standard Error of Mean 0.013 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration); Test type: Superiority; p < .0001, Mixed Models Analysis; Difference to Placebo = -7.12, 90% CI 2-sided [-9.41 to -4.78], Standard Error of Mean 0.015 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Cohort 1: PF-06882961 200 mg BID (1-week Titration); Test type: Superiority; p < .0001, Mixed Models Analysis; Difference to Placebo = -9.12, 90% CI 2-sided [-11.11 to -7.08], Standard Error of Mean 0.013 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration); Test type: Superiority; p < .0001, Mixed Models Analysis; Difference to Placebo = -7.18, 90% CI 2-sided [-9.32 to -4.99], Standard Error of Mean 0.014 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Cohort 3: Percent Change From Baseline in Body Weight at End of Treatment at Week 32
Description: Percent change from baseline in body weight at end of treatment was reported in this outcome measure. Analysis was performed using MMRM with treatment, time, strata (females versus males) and treatment-by-time interaction as fixed effects, natural log-transformed baseline as a covariate and the (natural log-transformed baseline)-by-time interaction with time fitted as a repeated effect and participant as a random effect. Values were back-transformed from the log scale. Percent change = 100*(back-transformed LS Mean - 1). Baseline was defined as the average of the duplicate measurements collected closest prior to dosing at Day 1.
Time Frame: Baseline, Week 32
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 19 | 37 | 37 | 36
Percent change | 1.40 (0.018) | -6.92 (0.014) | -7.15 (0.014) | -11.65 (0.014)
Statistical Analysis 1: Comparison: Cohort 3: Placebo vs Cohort 3: PF-06882961 80mg BID (4-week Titration); Test type: Superiority; p < .0001, Mixed Models Analysis; Difference to Placebo = -8.21, 90% CI 2-sided [-11.66 to -4.63], Standard Error of Mean 0.023 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 3: Placebo vs Cohort 3: PF-06882961 140mg BID (4-week Titration); Test type: Superiority; p < .0001, Mixed Models Analysis; Difference to placebo = -8.44, 90% CI 2-sided [-11.83 to -4.92], Standard Error of Mean 0.023 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort 3: Placebo vs Cohort 3: PF-06882961 200mg BID (4-week Titration); Test type: Superiority; p < .0001, Mixed Models Analysis; Difference to Placebo = -12.87, 90% CI 2-sided [-16.15 to -9.47], Standard Error of Mean 0.023 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Cohorts 1 and 2: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious AEs (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose met one or more of the criteria such as resulted in death; life threatening; required inpatient hospitalization or prolongation of existing hospitalization; persistent disability or incapacity, congenital anomaly or birth defect; suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic. An adverse event is considered treatment-emergent relative to given treatment if the event starts during the effective duration of the treatment (i.e. starting on or after the first dose but before the last dose plus follow-up period).
Time Frame: From first dose of study intervention on Day 1 up to 28-35 days after last dose of study treatment (maximum up to 31 weeks)
Population: Safety analysis set included all participants randomly assigned to study intervention of the study and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 71 | 62 | 63 | 64 | 38 | 63 | 37 | 63 | 36
Participants
  TEAEs | 50 | 52 | 59 | 54 | 32 | 59 | 30 | 59 | 30
  TESAEs | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 5 | 1

4. Secondary Outcome: Cohort 3: Number of Participants With TEAEs and TESAEs
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose met one or more of the criteria such as resulted in death; life threatening; required inpatient hospitalization or prolongation of existing hospitalization; persistent disability or incapacity, congenital anomaly or birth defect; suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic. An adverse event is considered treatment-emergent relative to given treatment if the event starts during the effective duration of the treatment (i.e. starting on or after the first dose but before the last dose plus lag time).
Time Frame: From first dose of study intervention on Day 1 up to 28-35 days after last dose of study treatment (maximum up to 37 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 19 | 37 | 37 | 36
Participants
  TEAEs | 13 | 30 | 34 | 34
  TESAEs | 0 | 2 | 2 | 3

5. Secondary Outcome: Cohorts 1 and 2: Number of Participants With Laboratory Abnormalities, Without Regard to Baseline Abnormality
Description: Laboratory parameters:a)hematology:hemoglobin(Hg),hematocrit,erythrocytes(ery),neutrophils,ery mean corpuscular volume,platelets,leukocytes(leu),lymphocytes,basophils,eosinophils,monocytes activated partial thromboplastin time, prothrombin time,prothrombin initial normalised ratio b)chemistry:direct bilirubin(bil),indirect bil, gamma glutamyl transferase,urea nitrogen,urate,sodium,potassium,calcium(cal),cal corrected,bicarbonate,Hg a1c,creatine kinase,bile acid,calcitonin,insulin-fasting,glucose fasting,amylase,lipase,thyrotropin,thyroxine,free,cholesterol,high density lipoprotein (hdl) cholesterol,triglycerides,alanine aminotransferase c)urinalysis:urine:pH,ketone,protein, Hg, urobilinogen,nitrite,leu esterase,ery,leu,tubular epithelial cells,squamous epithelial cells,granular casts,hyaline casts,uric acid crystals,calcium oxalate crystals,amorphous crystals,mucus,microscopic exam,spermatozoa,yeast budding,transitional epithelial cells,leu cell clumps;yeast hyphae.
Time Frame: From first dose of study intervention on Day 1 up to 28-35 days after last dose of study treatment (up to 31 weeks)
Population: Safety analysis set included all participants randomly assigned to study intervention of the study and who took at least 1 dose of study intervention. Here "Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 69 | 61 | 63 | 64 | 37 | 62 | 34 | 63 | 35
Participants | 66 | 56 | 60 | 57 | 37 | 54 | 33 | 59 | 33

6. Secondary Outcome: Cohort 3: Number of Participants With Laboratory Abnormalities, Without Regard to Baseline Abnormality
Description: as for outcome 5
Time Frame: From first dose of study intervention on Day 1 up to 28-35 days after last dose of study treatment (up to 37 weeks)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 17 | 35 | 37 | 34
Participants | 15 | 31 | 34 | 32

7. Secondary Outcome: Cohorts 1 and 2: Number of Participants According to Categorization of Vital Signs Data
Description: Vital signs of systolic blood pressure, diastolic blood pressure and pulse rate and were measured using an automated device with the participant in a supine position after five minutes of rest. This reports the number of participants that met the following pre-specified criteria: systolic blood pressure (SBP) <90 millimetres of mercury (mmHg), diastolic blood pressure (DBP) <50 mmHg, pulse rate (PR) <40 beats per minute, >120 beats per minute.
Time Frame: From first dose of study intervention on Day 1 up to 28-35 days after last dose of study treatment (up to 31 weeks)
Population: Safety analysis set included all participants randomly assigned to study intervention of the study and who took at least 1 dose of study intervention. Here "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 70 | 62 | 63 | 64 | 38 | 63 | 37 | 63 | 36
Participants
  SBP Value < 90 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0
  DBP Value < 50 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  PR <40 beats per minute | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR >120 beats per minute | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Cohort 3: Number of Participants According to Categorization of Vital Signs Data
Description: as for outcome 7
Time Frame: From first dose of study intervention on Day 1 up to 28-35 days after last dose of study treatment (up to 37 weeks)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 18 | 37 | 37 | 36
Participants
  DBP Value < 50 | 0 | 0 | 1 | 0
  SBP Value < 90 | 0 | 0 | 0 | 0
  PR <40 beats per minute | 0 | 0 | 0 | 0
  PR >120 beats per minute | 0 | 0 | 0 | 0

9. Secondary Outcome: Cohorts 1 and 2: Number of Participants According to Categorization of Electrocardiogram (ECG) Parameters
Description: Standard 12-lead ECGs were measured with the participant in a supine position after at least five minutes of rest. This reports the number of participants that met the following pre-specified criteria for ECG: QRS interval >=140; PR interval >=300; QTCF interval >500.
Time Frame: From first dose of study intervention on Day 1 up to 28-35 days after last dose of study treatment (up to 31 weeks)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 69 | 61 | 63 | 64 | 37 | 62 | 34 | 63 | 35
Participants
  QRS interval >=140 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  QTCF interval >500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR interval >=300 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Cohort 3: Number of Participants According to Categorization of ECG Parameters
Description: as for outcome 9
Time Frame: From first dose of study intervention on Day 1 up to 28-35 days after last dose of study treatment (up to 37 weeks)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 17 | 35 | 37 | 34
Participants
  QRS interval >=140 | 0 | 0 | 0 | 1
  QTCF interval >500 | 0 | 0 | 0 | 0
  PR interval >=300 | 0 | 0 | 0 | 0

11. Secondary Outcome: Cohorts 1 and 2: Number of Participants With Categorical Scores on Columbia-Suicide Severity Rating Scale (C-SSRS) Leading to Study Discontinuation
Description: C-SSRS is an interview-based rating scale to assess suicidal ideation and behavior. Per protocol, any participant with a pre-specified score was required to be evaluated by a mental health professional and, if meeting pre-defined criteria, discontinued from the study.
Time Frame: Week 0 (Baseline), 2, 4, 6, 8, 10, 12, 16, 18, 22, 26, Follow-up (Week 31)
Population: Safety analysis set included all participants randomly assigned to study intervention of the study and who took at least 1 dose of study intervention. Here, "Number of Participants analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 71 | 62 | 63 | 64 | 38 | 63 | 37 | 63 | 36
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Cohort 3: Number of Participants With Categorical Scores on C-SSRS Leading to Study Discontinuation
Description: as for outcome 11
Time Frame: Week 0 (Baseline), 4, 8, 12, 16, 20, 24, 28, 32, Follow-up (Week 37)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 19 | 37 | 37 | 36
Participants | 0 | 0 | 0 | 0

13. Secondary Outcome: Cohort 1 and 2: Number of Participants With Scores on the Patient Health Questionnaire-9 (PHQ-9) Leading to Study Discontinuation
Description: PHQ-9 is a self-reported, nine-item scale for the assessment of depressive disorder. Per protocol, any participant with a pre-specified score was required to be evaluated by a mental health professional and, if meeting pre-defined criteria, discontinued from the study.
Time Frame: Week 0 (Baseline) , 2, 4, 6, 8, 10, 12, 16, 18, 22, 26, Follow-up (Week 31)
Population: Safety analysis set included all participants randomly assigned to study intervention of the study and who took at least 1 dose of study intervention. Here, 'Number Analyzed' signifies participants evaluable for the specified rows."
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 71 | 62 | 63 | 64 | 38 | 63 | 37 | 63 | 36
Participants | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

14. Secondary Outcome: Cohort 3: Number of Participants With Scores on the PHQ-9 Leading to Study Discontinuation
Description: as for outcome 13
Time Frame: Week 0 (Baseline), 4, 8, 12, 16, 20, 24, 28, 32, Follow-up (Week 37)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 19 | 37 | 37 | 36
Participants | 0 (0) | 0 (0) | 0 (0) | 0 (0)

15. Secondary Outcome: Cohorts 1 and 2: Number of Participants With >= 5% Body Weight Loss at End of Treatment
Description: Number of participants with >= 5% body weight loss at end of treatment were reported.
Time Frame: Week 26
Population: Estimand Set 1 included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Here, "Number of Participants analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 44 | 27 | 30 | 26 | 14 | 18 | 11 | 14 | 13
Participants | 6 | 16 | 15 | 17 | 12 | 15 | 6 | 12 | 8
Statistical Analysis 1: Comparison: Cohorts 1 and 2: Placebo vs Cohort 1: PF-06882961 40mg BID (1-week Titration); Test type: Superiority — Logistic regression models (included terms for treatment, strata [females versus males] and baseline body weight as a covariate) were applied to the imputed datasets from the multiple imputation method above and parameter estimates were combined using standard multiple imputation techniques; Odds Ratio (OR) = 7.37, 90% CI 2-sided [2.81 to 19.30]
Statistical Analysis 2: Comparison: Cohorts 1 and 2: Placebo vs Cohort 1: PF-06882961 80mg BID (1-week Titration); Logistic regression models (included terms for treatment, strata [females versus males] and baseline body weight as a covariate) were applied to the imputed datasets from the multiple imputation method above and parameter estimates were combined using standard multiple imputation techniques; Test type: Superiority; Odds Ratio (OR) = 6.58, 90% CI 2-sided [2.62 to 16.53]
Statistical Analysis 3: Comparison: Cohorts 1 and 2: Placebo vs Cohort 1: PF-06882961 120mg BID (1-week Titration); [analysis description as in outcome 15, analysis 2]; Test type: Superiority; Odds Ratio (OR) = 16.33, 90% CI 2-sided [6.47 to 41.24]
Statistical Analysis 4: Comparison: Cohorts 1 and 2: Placebo vs Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration); Test type: Superiority — [test comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 14.24, 90% CI 2-sided [5.39 to 37.66]
Statistical Analysis 5: Comparison: Cohorts 1 and 2: Placebo vs Cohort 1: PF-06882961 160 mg BID (1-week Titration); Test type: Superiority — [test comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 30.17, 90% CI 2-sided [11.35 to 80.20]
Statistical Analysis 6: Comparison: Cohorts 1 and 2: Placebo vs Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration); Test type: Superiority — [test comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 9.88, 90% CI 2-sided [2.91 to 33.53]
Statistical Analysis 7: Comparison: Cohorts 1 and 2: Placebo vs Cohort 1: PF-06882961 200 mg BID (1-week Titration); Test type: Superiority — [test comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 24.41, 90% CI 2-sided [8.28 to 71.95]
Statistical Analysis 8: Comparison: Cohorts 1 and 2: Placebo vs Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration); Test type: Superiority — [test comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 12.65, 90% CI 2-sided [4.56 to 35.08]

16. Secondary Outcome: Cohort 3: Number of Participants With >=5% Body Weight Loss at End of Treatment
Description: Number of participants with >= 5% body weight loss at end of treatment were reported.
Time Frame: Week 32
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 11 | 13 | 15 | 11
Participants | 0 | 9 | 11 | 10
Statistical Analysis 1: Comparison: Cohort 3: Placebo vs Cohort 3: PF-06882961 80mg BID (4-week Titration); Test type: Superiority — [test comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 33.43, 90% CI 2-sided [3.05 to 366.64]
Statistical Analysis 2: Comparison: Cohort 3: Placebo vs Cohort 3: PF-06882961 140mg BID (4-week Titration); Test type: Superiority — [test comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 34.04, 90% CI 2-sided [3.10 to 373.85]
Statistical Analysis 3: Comparison: Cohort 3: Placebo vs Cohort 3: PF-06882961 200mg BID (4-week Titration); Test type: Superiority — [test comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 127.21, 90% CI 2-sided [10.55 to 1533.46]

17. Secondary Outcome: Cohorts 1 and 2: Percent Change From Baseline in Body Weight at Weeks 2, 4, 6, 8, 10, 12,16, 18, 22
Description: as for outcome 2
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12,16, 18, 22
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 71 | 62 | 63 | 64 | 38 | 63 | 37 | 63 | 36
Percent Change
  Week 2 | -0.13 (0.001) | -0.85 (0.001) | -0.54 (0.001) | -0.98 (0.001) | -0.58 (0.002) | -0.87 (0.001) | -0.22 (0.002) | -0.96 (0.001) | -0.53 (0.002)
  Week 4 | -0.15 (0.002) | -1.65 (0.002) | -1.69 (0.002) | -1.99 (0.002) | -1.26 (0.003) | -1.71 (0.002) | -0.93 (0.003) | -1.98 (0.002) | -1.28 (0.003)
  Week 6 | -0.24 (0.003) | -2.26 (0.003) | -2.37 (0.003) | -2.96 (0.003) | -1.99 (0.003) | -2.84 (0.003) | -1.93 (0.004) | -2.97 (0.003) | -1.99 (0.004)
  Week 8 | -0.41 (0.003) | -2.93 (0.003) | -2.86 (0.003) | -3.89 (0.003) | -3.33 (0.004) | -3.87 (0.004) | -2.34 (0.004) | -3.83 (0.004) | -2.94 (0.004)
  Week 10 | -0.50 (0.004) | -3.47 (0.004) | -3.33 (0.004) | -4.82 (0.004) | -3.92 (0.005) | -4.67 (0.004) | -3.20 (0.005) | -4.54 (0.004) | -3.83 (0.005)
  Week 12 | -0.44 (0.004) | -3.89 (0.005) | -3.88 (0.004) | -5.31 (0.005) | -4.49 (0.006) | -5.66 (0.005) | -3.98 (0.006) | -5.33 (0.005) | -4.34 (0.006)
  Week 16 | -0.40 (0.005) | -4.73 (0.006) | -4.01 (0.006) | -6.98 (0.006) | -5.49 (0.008) | -7.04 (0.007) | -5.15 (0.008) | -6.56 (0.007) | -5.18 (0.008)
  Week 18 | -0.50 (0.006) | -4.94 (0.006) | -4.68 (0.006) | -7.33 (0.007) | -6.33 (0.008) | -7.50 (0.007) | -5.57 (0.009) | -7.27 (0.007) | -5.80 (0.008)
  Week 22 | -0.18 (0.007) | -5.06 (0.008) | -5.00 (0.007) | -8.10 (0.008) | -6.43 (0.010) | -8.63 (0.009) | -6.57 (0.011) | -8.23 (0.009) | -6.60 (0.010)

18. Secondary Outcome: Cohort 3: Percent Change From Baseline in Body Weight at Weeks 4, 8, 12, 16, 20, 24 and 28
Description: as for outcome 2
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24 and 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 19 | 37 | 37 | 36
Percent Change
  Week 4 | -0.37 (0.004) | -1.38 (0.003) | -0.95 (0.003) | -1.02 (0.003)
  Week 8 | -0.06 (0.006) | -2.07 (0.004) | -1.93 (0.004) | -1.89 (0.004)
  Week 12 | -0.08 (0.008) | -2.80 (0.006) | -2.88 (0.005) | -2.96 (0.006)
  Week 16 | 0.03 (0.011) | -4.13 (0.008) | -3.99 (0.007) | -4.73 (0.008)
  Week 20 | 0.38 (0.014) | -5.17 (0.010) | -5.25 (0.009) | -7.10 (0.010)
  Week 24 | 0.36 (0.015) | -5.65 (0.011) | -6.39 (0.011) | -9.20 (0.011)
  Week 28 | 1.06 (0.017) | -6.37 (0.013) | -6.74 (0.012) | -10.44 (0.013)

19. Secondary Outcome: Cohorts 1 and 2: Absolute Change From Baseline in Waist Circumference at End of Treatment at Week 26
Description: Absolute change from baseline in waist circumference were reported. Analysis was performed using MMRM model with treatment, time, strata (females versus males) and treatment-by-time interaction as fixed effects, baseline as a covariate and the baseline-by-time interaction with time fitted as a repeated effect and participant as a random effect. Baseline was defined as the average of the duplicate measurements collected closest prior to dosing at Day 1.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Centimeter
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 71 | 62 | 63 | 64 | 38 | 63 | 37 | 63 | 36
Centimeter | -1.25 (0.826) | -6.49 (0.995) | -5.75 (0.943) | -6.19 (1.023) | -5.98 (1.338) | -9.05 (1.174) | -7.41 (1.490) | -7.56 (1.281) | -6.36 (1.350)

20. Secondary Outcome: Cohort 3: Absolute Change From Baseline in Waist Circumference at End of Treatment at Week 32
Description: as for outcome 19
Time Frame: Baseline, Week 32
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Centimeter
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 19 | 37 | 37 | 36
Centimeter | 0.19 (1.967) | -6.27 (1.628) | -7.77 (1.564) | -11.43 (1.698)

21. Secondary Outcome: Cohorts 1 and 2: Absolute Change From Baseline in Waist-to-hip Ratio at End of Treatment at Week 26
Description: Absolute change from baseline in waist-to-hip ratio at end of treatment were reported. Analysis was performed using MMRM model with treatment, time, strata (females versus males) and treatment-by-time interaction as fixed effects, baseline as a covariate and the baseline-by-time interaction with time fitted as a repeated effect and participant as a random effect. Baseline was defined as the average of the duplicate measurements collected closest prior to dosing at Day 1.
Time Frame: Baseline, Week 26
Population: Estimand Set 1 included all participants randomly assigned to study intervention in Part A and who took at least 1 dose of study intervention.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 71 | 62 | 63 | 64 | 38 | 63 | 37 | 63 | 36
Ratio | -0.002 (0.0064) | -0.002 (0.0076) | -0.015 (0.0073) | 0.001 (0.0078) | -0.014 (0.0104) | -0.015 (0.0090) | -0.014 (0.0114) | -0.007 (0.0098) | 0.004 (0.0104)

22. Secondary Outcome: Cohort 3: Absolute Change From Baseline in Waist-to-hip Ratio at End of Treatment at Week 32
Description: as for outcome 21
Time Frame: Baseline, Week 32
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 19 | 37 | 37 | 36
Ratio | 0.010 (0.0128) | -0.012 (0.0113) | -0.009 (0.0108) | -0.016 (0.0121)

23. Secondary Outcome: Cohorts 1 and 2: Absolute Change From Baseline in Percentage Hemoglobin A1c (HbA1c) at Weeks 16 and 26
Description: Absolute change from baseline in HbA1c were reported. Analysis was performed using MMRM model with treatment, time, strata (females versus males) and treatment-by-time interaction as fixed effects, baseline as a covariate and the baseline-by-time interaction with time fitted as a repeated effect and participant as a random effect. Baseline was defined as the average of the duplicate measurements collected closest prior to dosing at Day 1.
Time Frame: Baseline, Weeks 16 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 71 | 62 | 63 | 64 | 38 | 63 | 37 | 63 | 36
Percentage of HbA1c
  Week 16 | 0.00 (0.034) | -0.24 (0.039) | -0.24 (0.039) | -0.26 (0.042) | -0.25 (0.056) | -0.29 (0.050) | -0.18 (0.061) | -0.23 (0.053) | -0.24 (0.054)
  Week 26 | 0.01 (0.036) | -0.17 (0.045) | -0.13 (0.044) | -0.22 (0.046) | -0.16 (0.064) | -0.31 (0.055) | -0.13 (0.070) | -0.17 (0.062) | -0.26 (0.064)

24. Secondary Outcome: Cohort 3: Absolute Change From Baseline in Percentage HbA1c at Weeks 16, 24 and 32
Description: as for outcome 23
Time Frame: Baseline, Weeks 16, 24 and 32
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 19 | 37 | 37 | 36
Percentage of HbA1c
  Week 16 | -0.05 (0.061) | -0.16 (0.048) | -0.26 (0.044) | -0.29 (0.042)
  Week 24 | 0.05 (0.070) | -0.13 (0.059) | -0.21 (0.055) | -0.31 (0.059)
  Week 32 | -0.02 (0.074) | -0.11 (0.064) | -0.27 (0.059) | -0.41 (0.068)

25. Secondary Outcome: Cohorts 1 and 2: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) at Weeks 2, 4, 6, 8, 10, 12, 16, 18, 22, 26
Description: Absolute change from baseline in FPG were reported. Analysis was performed using MMRM model with treatment, time, strata (females versus males) and treatment-by-time interaction as fixed effects, baseline as a covariate and the baseline-by-time interaction with time fitted as a repeated effect and participant as a random effect. Baseline was defined as the average of the duplicate measurements collected closest prior to dosing at Day 1.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 16, 18, 22, 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Milligram per deciliter
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration)
Number analyzed (Participants) | 71 | 62 | 63 | 64 | 38 | 63 | 37 | 63 | 36
Milligram per deciliter
  Week 2 | 3.22 (0.903) | -2.93 (0.963) | -2.56 (0.939) | -4.02 (0.940) | -2.02 (1.245) | -4.51 (0.957) | -1.16 (1.265) | -2.82 (0.939) | -2.93 (1.250)
  Week 4 | 3.38 (1.082) | -2.75 (1.196) | -2.97 (1.166) | -3.59 (1.155) | -0.83 (1.443) | -4.81 (1.199) | -2.56 (1.504) | -6.24 (1.164) | -3.86 (1.485)
  Week 6 | 1.45 (0.936) | -4.28 (1.021) | -2.29 (1.035) | -6.38 (1.044) | -4.17 (1.290) | -3.46 (1.102) | -3.06 (1.371) | -4.32 (1.095) | -4.64 (1.311)
  Week 8 | 1.61 (0.956) | -3.72 (1.068) | -3.15 (1.103) | -2.56 (1.130) | -2.77 (1.385) | -4.48 (1.177) | -4.07 (1.438) | -4.90 (1.248) | -2.82 (1.367)
  Week 10 | 2.47 (1.146) | -2.52 (1.264) | -1.79 (1.251) | -4.74 (1.353) | -2.60 (1.662) | -4.17 (1.498) | -5.26 (1.702) | -5.35 (1.525) | -2.85 (1.558)
  Week 12 | 2.57 (1.229) | -2.70 (1.408) | -0.77 (1.377) | -2.24 (1.492) | -1.22 (1.889) | -4.86 (1.686) | -4.65 (1.908) | -3.01 (1.716) | -3.19 (1.764)
  Week 16 | 0.50 (1.352) | -2.67 (1.523) | -2.04 (1.537) | -2.56 (1.619) | -6.99 (2.143) | -6.62 (1.926) | -5.73 (2.338) | -4.67 (2.011) | -5.24 (2.097)
  Week 18 | 4.34 (1.407) | -0.44 (1.634) | -3.73 (1.593) | 0.19 (1.770) | -0.96 (2.294) | -4.76 (2.030) | -5.23 (2.684) | 0.11 (2.175) | 0.53 (2.189)
  Week 22 | 4.83 (1.494) | 0.38 (1.872) | -3.22 (1.712) | -4.27 (1.842) | -1.78 (2.502) | -2.03 (2.205) | -1.65 (2.888) | -4.64 (2.460) | -5.08 (2.580)
  Week 26 | 3.34 (1.220) | -3.37 (1.499) | -3.43 (1.469) | -4.02 (1.555) | -3.75 (2.059) | -6.00 (1.804) | -3.50 (2.290) | -6.60 (2.010) | -5.01 (2.172)

26. Secondary Outcome: Cohort 3: Absolute Change From Baseline in FPG at Weeks 4, 8, 12, 16, 20, 24, 28, 32
Description: as for outcome 25
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Milligram per deciliter
Arm/Group | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
Number analyzed (Participants) | 19 | 37 | 37 | 36
Milligram per deciliter
  Week 4 | -1.82 (2.327) | -0.83 (1.652) | 0.96 (1.616) | 3.84 (1.671)
  Week 8 | 0.10 (2.523) | 1.79 (1.748) | -1.16 (1.659) | 2.52 (1.720)
  Week 12 | -1.28 (2.588) | -1.80 (1.883) | 1.56 (1.755) | -0.42 (1.761)
  Week 16 | -5.75 (2.348) | -5.18 (1.778) | -2.43 (1.654) | 0.88 (1.618)
  Week 20 | 1.52 (2.175) | -1.95 (1.774) | -4.78 (1.687) | -1.39 (1.628)
  Week 24 | -2.80 (2.664) | -0.13 (2.088) | -2.00 (2.014) | 1.62 (2.158)
  Week 28 | 1.67 (2.518) | -0.15 (2.044) | -4.53 (1.983) | 0.90 (2.221)
  Week 32 | -1.81 (3.006) | 1.28 (2.491) | -1.65 (2.446) | -1.73 (2.582)

ADVERSE EVENTS:
Time Frame: From first dose of study intervention on Day 1 up to 28-35 days after last dose of study treatment (maximum up to Week 31 for Cohort 1 and 2; maximum up to Week 37 for Cohort 3)
Description: An AE was any untoward medical occurrence in a participant temporally associated with use of study intervention, whether or not considered related to study intervention. Same event may appear as both non-SAE and SAE; however, what is presented are distinct events. Event may be categorized as serious in 1 participant and non-serious in another or may have experienced both SAE and non-SAE. All-causality non-SAEs occurring in >=5% of participants in any treatment group are included below.
Arm/Group | Cohorts 1 and 2: Placebo | Cohort 1: PF-06882961 40 mg BID (1-week Titration) | Cohort 1: PF-06882961 80mg BID (1-week Titration) | Cohort 1: PF-06882961 120mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration) | Cohort 3: Placebo | Cohort 3: PF-06882961 80mg BID (4-week Titration) | Cohort 3: PF-06882961 140mg BID (4-week Titration) | Cohort 3: PF-06882961 200mg BID (4-week Titration)
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/62 | 0/63 | 0/64 | 0/38 | 0/63 | 0/37 | 0/63 | 0/36 | 0/19 | 0/37 | 0/37 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/71 | 2/62 | 1/63 | 0/64 | 1/38 | 1/63 | 0/37 | 5/63 | 1/36 | 0/19 | 2/37 | 2/37 | 3/36
Other Adverse Events (participants affected / at risk) | 29/71 | 46/62 | 53/63 | 51/64 | 31/38 | 56/63 | 29/37 | 56/63 | 26/36 | 13/19 | 28/37 | 33/37 | 34/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohorts 1 and 2: Placebo (N=71) | Cohort 1: PF-06882961 40 mg BID (1-week Titration) (N=62) | Cohort 1: PF-06882961 80mg BID (1-week Titration) (N=63) | Cohort 1: PF-06882961 120mg BID (1-week Titration) (N=64) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) (N=38) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) (N=63) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) (N=37) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) (N=63) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration) (N=36) | Cohort 3: Placebo (N=19) | Cohort 3: PF-06882961 80mg BID (4-week Titration) (N=37) | Cohort 3: PF-06882961 140mg BID (4-week Titration) (N=37) | Cohort 3: PF-06882961 200mg BID (4-week Titration) (N=36)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohorts 1 and 2: Placebo (N=71) | Cohort 1: PF-06882961 40 mg BID (1-week Titration) (N=62) | Cohort 1: PF-06882961 80mg BID (1-week Titration) (N=63) | Cohort 1: PF-06882961 120mg BID (1-week Titration) (N=64) | Cohorts 1 and 2: PF-06882961 120 mg BID (2-week Titration) (N=38) | Cohort 1: PF-06882961 160 mg BID (1-week Titration) (N=63) | Cohorts 1 and 2: PF-06882961 160 mg BID (2-week Titration) (N=37) | Cohort 1: PF-06882961 200 mg BID (1-week Titration) (N=63) | Cohorts 1 and 2: PF-06882961 200 mg BID (2-week Titration) (N=36) | Cohort 3: Placebo (N=19) | Cohort 3: PF-06882961 80mg BID (4-week Titration) (N=37) | Cohort 3: PF-06882961 140mg BID (4-week Titration) (N=37) | Cohort 3: PF-06882961 200mg BID (4-week Titration) (N=36)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 4 | 2 | 0 | 1 | 3 | 0 | 5 | 1 | 0 | 2 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 3 | 3 | 3 | 5 | 2 | 3 | 2 | 0 | 1 | 2 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 5 | 2 | 3 | 6 | 1 | 1 | 0 | 1 | 3 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 | 2 | 6 | 1 | 3 | 1 | 5 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 8 | 10 | 7 | 5 | 12 | 4 | 9 | 6 | 2 | 7 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 7 | 5 | 17 | 12 | 9 | 13 | 3 | 11 | 6 | 1 | 8 | 8 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 6 | 11 | 5 | 5 | 13 | 2 | 13 | 4 | 1 | 5 | 3 | 7
Eructation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 4 | 0 | 0 | 2 | 3 | 1
Flatulence (Gastrointestinal disorders) | 1 | 4 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 7 | 8 | 8 | 10 | 3 | 4 | 10 | 6 | 1 | 2 | 2 | 8
Nausea (Gastrointestinal disorders) | 11 | 28 | 39 | 41 | 22 | 36 | 25 | 34 | 18 | 2 | 14 | 27 | 25
Vomiting (Gastrointestinal disorders) | 2 | 10 | 24 | 26 | 16 | 27 | 11 | 29 | 16 | 1 | 3 | 14 | 17
Chills (General disorders) | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 3 | 4 | 7 | 0 | 6 | 5 | 7 | 2 | 1 | 5 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 4 | 8 | 4 | 1 | 3 | 0 | 4 | 2 | 0 | 4 | 3 | 5
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 3 | 3 | 0 | 1 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 6 | 4 | 1 | 4 | 0 | 2 | 0 | 0 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 4 | 1 | 5 | 2 | 4 | 2 | 6 | 0 | 0 | 1 | 3 | 1
Headache (Nervous system disorders) | 8 | 6 | 11 | 11 | 3 | 11 | 6 | 7 | 6 | 3 | 5 | 3 | 4
Tremor (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 3 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Prehypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT04707313/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT04707313/SAP_001.pdf